CLINICAL TRIAL: NCT00152022
Title: A Phase III, Randomized, Double-blind, Multi-center, Placebo-controlled, Parallel-Group, Safety and Efficacy Study of SPD465 in Adults With Attention-Deficit Hyperactivity Disorder (ADHD).
Brief Title: Efficacy and Safety of SPD465 in Adults With Moderately Symptomatic ADHD.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SPD465-303
Record Dates: First submitted 2005-09-07; First posted 2005-09-09 (Estimated); Last update posted 2021-07-13 (Actual); Status verified 2021-07

CONDITIONS: Attention Deficit Disorder With Hyperactivity
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Amphetamine; Fumigant 93

INTERVENTIONS:
Drug: Neutral salts of dextroamphetamine sulfate, USP, amphetamine sulphate, USP, d-amphetamine saccharate, d, l-amphetamine aspartate monohydrate.

SUMMARY:
The purpose of this study is to assess the safety and effectiveness of SPD465 compared to placebo (a capsule with no medication in it) in the treatment of ADHD. The study will also look at how SPD465 affects the participants sleep and how they perceive their quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Primary diagnosis of ADHD
* Baseline ADHD-RS-IV score >= 32
* Non-pregnant females of childbearing potential must comply with contraceptive restrictions.

Exclusion Criteria:

* Significantly underweight or morbidly obese
* Comorbid psychiatric diagnosis with significant symptoms such as Axis II disorders or severe Axis I disorders
* History of seizure, tic disorder, or a current diagnosis and/or family history of Tourette's Disorder
* Females who are pregnant or lactating

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 412
Dates: Start 2005-04-25 (Actual); Primary Completion 2005-11-04 (Actual); Study Completion 2005-11-04 (Actual)

PRIMARY OUTCOMES:
The primary measure of efficacy will be the clinician-administered ADHD-rating scale (ADHD-RS-IV) | Baseline (following ADHD medication washout of 7-28 days)
  The ADHD-RS-IV consists of 18 items designed to reflect current symptomatology of ADHD. Each item is scored on a 4-point scale ranging from 0 (no symptoms) to three (severe symptoms), with the total score for the rating scale ranging from 0 to 54.
The primary measure of efficacy will be the clinician-administered ADHD-rating scale (ADHD-RS-IV) | Week 1
  The ADHD-RS-IV consists of 18 items designed to reflect current symptomatology of ADHD. Each item is scored on a 4-point scale ranging from 0 (no symptoms) to three (severe symptoms), with the total score for the rating scale ranging from 0 to 54.
The primary measure of efficacy will be the clinician-administered ADHD-rating scale (ADHD-RS-IV) | Week 2
  The ADHD-RS-IV consists of 18 items designed to reflect current symptomatology of ADHD. Each item is scored on a 4-point scale ranging from 0 (no symptoms) to three (severe symptoms), with the total score for the rating scale ranging from 0 to 54.
The primary measure of efficacy will be the clinician-administered ADHD-rating scale (ADHD-RS-IV) | Week 3
  The ADHD-RS-IV consists of 18 items designed to reflect current symptomatology of ADHD. Each item is scored on a 4-point scale ranging from 0 (no symptoms) to three (severe symptoms), with the total score for the rating scale ranging from 0 to 54.
The primary measure of efficacy will be the clinician-administered ADHD-rating scale (ADHD-RS-IV) | Week 4
  The ADHD-RS-IV consists of 18 items designed to reflect current symptomatology of ADHD. Each item is scored on a 4-point scale ranging from 0 (no symptoms) to three (severe symptoms), with the total score for the rating scale ranging from 0 to 54.
The primary measure of efficacy will be the clinician-administered ADHD-rating scale (ADHD-RS-IV) | Week 5
  The ADHD-RS-IV consists of 18 items designed to reflect current symptomatology of ADHD. Each item is scored on a 4-point scale ranging from 0 (no symptoms) to three (severe symptoms), with the total score for the rating scale ranging from 0 to 54.
The primary measure of efficacy will be the clinician-administered ADHD-rating scale (ADHD-RS-IV) | Week 6
  The ADHD-RS-IV consists of 18 items designed to reflect current symptomatology of ADHD. Each item is scored on a 4-point scale ranging from 0 (no symptoms) to three (severe symptoms), with the total score for the rating scale ranging from 0 to 54.

SECONDARY OUTCOMES:
Clinical Global Impression of Improvement scale (CG(-I) - assessed at visits 1 through 6/Early Termination (ET) | Weeks 1, 2, 3, 4, 5, & 6
Brown ADD Scale (BADDS) - completed at Baseline and 6/ET visits | Baseline visit and weeks 1, 2, 3, 4, 5, & 6
Adult ADHD Impact Module (AIM-A)-completed at Baseline and 6/ET visits. | Baseline visit and weeks 1, 2, 3, 4, 5, & 6
Pittsburgh Sleep Quality Index (PSQI) - taken at every visit from Baseline to study completion. | Baseline visit and weeks 1, 2, 3, 4, 5, & 6

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda

REFERENCES:
- [Derived] Surman CB, Roth T. Impact of stimulant pharmacotherapy on sleep quality: post hoc analyses of 2 large, double-blind, randomized, placebo-controlled trials. J Clin Psychiatry. 2011 Jul;72(7):903-8. doi: 10.4088/JCP.11m06838. PMID 21824454
- [Derived] Brown TE, Landgraf JM. Improvements in executive function correlate with enhanced performance and functioning and health-related quality of life: evidence from 2 large, double-blind, randomized, placebo-controlled trials in ADHD. Postgrad Med. 2010 Sep;122(5):42-51. doi: 10.3810/pgm.2010.09.2200. PMID 20861587